CLINICAL TRIAL: NCT05976568
Title: A Phase II/III, Randomized, Open-label, Multi-center Study to Evaluate the Efficacy and Safety of QL1706 in Combination With Bevacizumab and/or Chemotherapy Versus Sintilimab in Combination With Bevacizumab as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of QL1706 in Combination With Bevacizumab and/or Chemotherapy as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-308
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; Oxaliplatin; Capecitabine; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): QL1706 in combination with bevacizumab and chemotherapy
  Interventions: Drug: QL1706; Drug: Bevacizumab; Drug: Oxaliplatin injection; Drug: Capecitabine
- Arm 2 (Experimental): QL1706 in combination with bevacizumab
  Interventions: Drug: QL1706; Drug: Bevacizumab
- Arm 3 (Experimental): QL1706 in combination with chemotherapy
  Interventions: Drug: QL1706; Drug: Oxaliplatin injection; Drug: Capecitabine
- Arm 4 (Active Comparator): Sintilimab in combination with bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Sintilimab

INTERVENTIONS:
Drug: QL1706 — 7.5 mg/kg administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 1; Arm 2; Arm 3
Drug: Bevacizumab — 15 mg/kg administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 1; Arm 2; Arm 4
Drug: Oxaliplatin injection — 85 mg/m2 administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 1; Arm 3
Drug: Capecitabine — 1000 mg/m2 orally twice daily for 14 days continuous dosing followed by a 7-day break of each 21-day cycle
  Arms: Arm 1; Arm 3
Drug: Sintilimab — 200 mg administered as IV infusion on Day 1 of each 21-day cycle
  Arms: Arm 4

SUMMARY:
The purpose of this study is to assess the efficacy and safety of QL1706 in combination with bevacizumab and/or chemotherapy versus sintilimab in combination with bevacizumab as first-line treatment in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate voluntarily and sign informed consent.
2. Age ≥ 18 and ≤ 80 years old, male or female.
3. Histological or cytological or clinical diagnosis of HCC
4. Barcelona Clinic Liver Cancer stage C. BCLC stage B, not suitable for radical surgery and/or local treatment.
5. No prior systemic therapy for HCC.
6. Child-Pugh ≤7 , no history of hepatic encephalopathy.

Exclusion Criteria:

1. Histologically or cytologically documented fibrolamellar hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, cholangiocarcinoma, etc.
2. History of malignancy other than HCC within 5 years prior to the start of study treatment.
3. History of liver transplantation, or planned to receive liver transplantation.
4. Moderate or severe ascites with clinical symptoms that require drainage, uncontrolled or moderate or severe pleural and pericardical effusion.
5. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
6. Involvement of both the main portal vein and the left and right branches by portal vein tumor thrombus, or of both the main trunk and the superior mesenteric vein concurrently, or of inferior vena cava.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (Phase II) | Up to approximately 4 years
  ORR was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Incidence of Adverse Events (AEs) (Phase II) | Up to approximately 4 years
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Overall Survival (OS) (Phase III) | Up to approximately 4 years
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 4 years
  ORR was assessed by investigators per RECIST 1.1
Disease Control Rate (DCR) | Up to approximately 4 years
  DCR was assessed by investigators per RECIST 1.1
Duration of Response (DOR) | Up to approximately 4 years
  DOR was assessed by investigators per RECIST 1.1
Progression-free Survival (PFS) | Up to approximately 4 years
  PFS was assessed by investigators per RECIST 1.1
Time to progression (TTP) | Up to approximately 4 years
  TTP was assessed by investigators per RECIST 1.1
Objective Response Rate (ORR) | Up to approximately 4 years
  ORR was assessed by investigators per mRECIST
Disease Control Rate (DCR) | Up to approximately 4 years
  DCR was assessed by investigators per mRECIST
Duration of Response (DOR) | Up to approximately 4 years
  DOR was assessed by investigators per mRECIST
Progression-free Survival (PFS) | Up to approximately 4 years
  PFS was assessed by investigators per mRECIST
Time to progression (TTP) | Up to approximately 4 years
  TTP was assessed by investigators per mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Fudan University; Shukui Qin, Principal Investigator — Nanjing Tianyinshan Hospital
Locations (2):
- China (2):
  - Nanjing Tianyinshan Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No